CLINICAL TRIAL: NCT02685163
Title: Natural Antioxidant Ice-cream Acutely Reduces Oxidative Stress, Improves Vascular Function and Physical Performance in Healthy Subjects
Brief Title: Natural Antioxidant Ice-cream, Oxidative Stress and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Davide Francomano, PhD Researcher, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Rif: 3727, Prot: 2325/15
Record Dates: First submitted 2016-02-08; First posted 2016-02-18 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Vascular System Injuries
MeSH Terms: conditions — Vascular System Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antioxidant Ice-cream (Experimental): Natural antioxidant Ice-cream
  Interventions: Other: Antioxidant ice-cream
- Control Ice-cream (Placebo Comparator): Natural control ice-cream
  Interventions: Other: Control Ice-cream

INTERVENTIONS:
Other: Antioxidant ice-cream — Narutal Antioxidant ice-cream
  Arms: Antioxidant Ice-cream
Other: Control Ice-cream — Natural Control Ice-cream
  Arms: Control Ice-cream

SUMMARY:
Formation of reactive oxygen species (ROS) contributes to pathogenesis and progression of several diseases. Polyphenols, have been shown to be beneficial against ROS.

This study evaluate the effects of a natural antioxidant ice-cream,rich in polyphenols, on oxidative stress, vascular function and physical performance. In this controlled, single-blind cross-over study, 14 healthy subjects were randomized to assume 100 mg of antioxidant ice-cream consisting of dark cocoa powder, extract of hazelnut and green tea, or milk chocolate ice-cream (control ice-cream). Subjects were studied at baseline and two hours after the ingestion of the ice-creams. Serum polyphenols, antioxidant status (ferric reducing ability of plasma, FRAP), NO bioavailability (NOx), markers of oxidative stress (D-Roms and H2O2), endothelium function (FMD and RHI) and exercise tolerance (Stress Test) with measurement of the double product were assessed.

DETAILED DESCRIPTION:
14 healthy, non-smoking, volunteers (7 males ), aged between 20 and 40 years were enrolled. The study was randomized, placebo-controlled. After enrollment, 3 days before entering the study, all subjects performed an exercise stress test. They were then randomly allocated to the treatment sequence with 100 mg of natural anti-oxidant ice cream or milk chocolate ice-cream (control icecream) in a cross-over single-blind design. There was 1 week wash-out between 2 phases of the study.

Markers of oxidative stress (D-ROMs and H2O2); serum antioxidant status (FRAP), NO bioavailability (NOx), the endothelium flow-mediated vasodilation (FMD and the RHI by Endopat 2000) were evaluated in fasting condition at baseline (time 0) and 2 hours after the ingestion of the anti-oxidant or control ice-creams. The exercise stress test was performed before randomization and 2 hours after each ice-cream meal test. In both experiments, the ice-cream was consumed within 10 min.

Each subject was asked to refrain from any kind of medication, diet integrators, intensive physical activity and to avoid consumption of polyphenols rich foods, such cocoa-containing products, red wine, tea within the previously 2 weeks. All participants gave written informed consent, and the study was approved by the Medical Ethics Committee of La Sapienza University of Rome (Rif: 3727, Prot: 2325/15).

ELIGIBILITY:
Inclusion Criteria:

* healthy, non-smoking, volunteers

Exclusion Criteria:

* Assumption of any kind of medication, diet integrators, intensive physical activity and to avoid consumption of polyphenols rich foods, tea within the previously 2 weeks.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Acute 2 hours
  Endothelial function will be performed By Endopat2000 and FMD

CONTACTS AND LOCATIONS:
Overall Officials: Davide Francomano, MD, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hooper L, Kroon PA, Rimm EB, Cohn JS, Harvey I, Le Cornu KA, Ryder JJ, Hall WL, Cassidy A. Flavonoids, flavonoid-rich foods, and cardiovascular risk: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2008 Jul;88(1):38-50. doi: 10.1093/ajcn/88.1.38. PMID 18614722